CLINICAL TRIAL: NCT01283373
Title: A Phase I, Open-Label Study of the Safety and Pharmacokinetics of Escalating Doses of DSTP3086S in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of the Safety and Pharmacokinetics of Escalating Doses of DSTP3086S in Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DST4964g; GO00768 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

ARMS (2):
- A (Experimental): Dose escalation cohorts
  Interventions: Drug: DSTP3086S
- B (Experimental): Dose expansion cohorts
  Interventions: Drug: DSTP3086S

INTERVENTIONS:
Drug: DSTP3086S — DSTP3086S administered intravenously
  Arms: B
Drug: DSTP3086S — Escalating intravenous dose
  Arms: A

SUMMARY:
This is a Phase I, multicenter, open-label, dose-escalation study of DSTP3086S administered as a single agent by intravenous (IV) infusion to patients with metastatic Castration-Resistant Prostate Cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* Histologic documentation of adenocarcinoma of the prostate
* Surgical castration or ongoing use of gonadotropin-releasing hormone agonists with confirmed castrate levels of testosterone
* Metastatic progressive CRPC defined as progressive disease despite surgical castration or ongoing use of gonadotropin-releasing hormone agonists with confirmed castrate levels of testosterone
* For patients in the dose-expansion cohort of the study, not more than two prior lines of cytotoxic chemotherapy in the metastatic setting
* Evaluable or measurable disease
* Documented willingness to use an effective means of contraception

Exclusion Criteria:

* Anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy, or radiotherapy within 4 weeks prior to Day 1, with the following exceptions: maintenance hormonal therapy for metastatic prostate cancer and palliative radiation to bone metastases within 2 weeks prior to Day 1
* Major surgical procedure within 4 weeks prior to Day 1
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including HIV and atypical mycobacterial disease, but excluding fungal infections of the nail beds)
* Ongoing corticosteroid use with > 10 mg of daily prednisone or equivalent
* Symptomatic hypercalcemia requiring continued use of bisphosphonate therapy. Patients who are receiving bisphosphonate therapy specifically to prevent skeletal events and who do not have a history of clinically significant hypercalcemia are eligible.
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Untreated or active central nervous system (CNS) metastases. Patients with a history of treated CNS metastases are eligible, provided that they meet all of the following criteria: evaluable or measurable disease outside the CNS, radiographic demonstration of improvement upon the completion of CNS-directed therapy and no evidence of interim progression between the completion of CNS-directed therapy and the screening radiographic study, and screening CNS radiographic study is >/= 8 weeks since completion of radiotherapy and >/= 4 weeks since the discontinuation of corticosteroids and anticonvulsants
* Dose expansion cohort (B): no prior chemotherapy is allowed

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of dose-limiting toxicities (DLTs) | Days 1-21

SECONDARY OUTCOMES:
Area under the concentration-time curve | Up to 1 year
Maximum and minimum concentrations | Up to 1 year
Clearance | Up to 1 year
Half-life | Up to 1 year
Volume of distribution | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Fine, M.D., Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - San Francisco, California
  - Chicago, Illinois
  - Detroit, Michigan
  - New York, New York
  - Seattle, Washington

REFERENCES:
- [Derived] Martiniova L, Zielinski RJ, Lin M, DePalatis L, Ravizzini GC. The Role of Radiolabeled Monoclonal Antibodies in Cancer Imaging and ADC Treatment. Cancer J. 2022 Nov-Dec 01;28(6):446-453. doi: 10.1097/PPO.0000000000000625. PMID 36383907
- [Derived] Danila DC, Szmulewitz RZ, Vaishampayan U, Higano CS, Baron AD, Gilbert HN, Brunstein F, Milojic-Blair M, Wang B, Kabbarah O, Mamounas M, Fine BM, Maslyar DJ, Ungewickell A, Scher HI. Phase I Study of DSTP3086S, an Antibody-Drug Conjugate Targeting Six-Transmembrane Epithelial Antigen of Prostate 1, in Metastatic Castration-Resistant Prostate Cancer. J Clin Oncol. 2019 Dec 20;37(36):3518-3527. doi: 10.1200/JCO.19.00646. Epub 2019 Nov 5. PMID 31689155